CLINICAL TRIAL: NCT07182656
Title: A Phase I Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Pharmacodynamics of Single and Multiple Doses of CIGB-814 in Healthy Participants
Brief Title: Safety, Tolerability, and PK/PD of CIGB-814 in Chinese Health Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yi Fang (Other)
Responsible Party: Sponsor-Investigator, Yi Fang, Professor of Pharmacy, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDLK-20250425PK-CIGB814
Record Dates: First submitted 2025-08-26; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CIGB-814 (single-dose group) (Experimental)
  Interventions: Drug: CIGB-814 (single-dose group)
- CIGB-814 placebo (single-dose group) (Placebo Comparator)
  Interventions: Drug: CIGB-814 placebo (single-dose group)
- CIGB-814 (multiple-dose group) (Experimental)
  Interventions: Drug: CIGB-814 (multiple-dose group)
- CIGB-814 placebo (multiple-dose group) (Placebo Comparator)
  Interventions: Drug: CIGB-814 placebo (multiple-dose group)

INTERVENTIONS:
Drug: CIGB-814 (single-dose group) — CIGB-814, single ascending dose, SC injection
  Arms: CIGB-814 (single-dose group)
Drug: CIGB-814 placebo (single-dose group) — CIGB-814 placebo, single ascending dose, SC injection
  Arms: CIGB-814 placebo (single-dose group)
Drug: CIGB-814 (multiple-dose group) — CIGB-814, multiple ascending dose, SC injection
  Arms: CIGB-814 (multiple-dose group)
Drug: CIGB-814 placebo (multiple-dose group) — CIGB-814 placebo, multiple ascending dose, SC injection
  Arms: CIGB-814 placebo (multiple-dose group)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of CIGB-814 for injection after single and multiple administrations in healthy participants. Secondary objectives include the assessment of preliminary pharmacodynamics (PD) and immunogenicity. Exploratory objectives are to investigate changes in immune cell subsets and signaling pathways following multiple administrations of CIGB-814.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be eligible for the study:

  1. Healthy male or female participants aged 18 to 45 years, inclusive.
  2. Male participants weighing at least 50.0 kg, and female participants weighing at least 45.0 kg, with a body mass index (BMI) between 19.0 and 26.0 kg/m², inclusive (BMI = weight [kg] / height² [m²]).
  3. Able to communicate effectively with the investigators, understand and comply with all study requirements, and willing to adhere strictly to the study procedures and follow-up schedule. Participants must provide written informed consent prior to any study-related procedures.
  4. From the date of signing the informed consent until 6 months after study completion, participants must not have plans for conception. Female participants must not have plans to donate oocytes and agree to use reliable contraception to avoid pregnancy. Male participants must not have plans to donate sperm and agree to use reliable contraception to prevent pregnancy of their partner.

Exclusion Criteria:

* Participants meeting any of the following criteria will be excluded from the study:

  1.History or presence of any clinically significant disease, including but not limited to:
  1. Respiratory (e.g., past or active tuberculosis), cardiovascular, gastrointestinal, urinary, musculoskeletal, endocrine (e.g., adrenal insufficiency), neurological or psychiatric (e.g., epilepsy), hematologic (particularly any hemolytic disorders such as glucose-6-phosphate dehydrogenase [G6PD] deficiency or paroxysmal nocturnal hemoglobinuria [PNH]), immune system disorders, or known significant bleeding tendencies;
  2. Fever or infectious disease within 3 days prior to screening;
  3. History of gastrointestinal, liver, or kidney diseases, including prior partial resection of these organs;
  4. Severe infection, trauma, or surgery within 12 weeks prior to screening, or planned surgery during the study deemed unsuitable by the investigator;
  5. Clinically significant acute illness (e.g., gastrointestinal disorders, infections) within 4 weeks prior to screening;
  6. Chronic pain (persistent or recurrent for >3 months) or currently experiencing acute pain (<3 months).

  2.History of significant allergies, including known hypersensitivity to any investigational product or its components, food allergies, pollen allergies, or other allergic conditions.

  3.Smoking more than 5 cigarettes per day (or equivalent tobacco use) within 3 months prior to screening, or inability to abstain from tobacco during the study.

  4.History of alcohol abuse, average alcohol consumption ≥14 units/week within 3 months prior to screening (1 unit = 10 mL ethanol, e.g., 200 mL beer [5%], 25 mL spirits [40%], or 83 mL wine [12%]), positive alcohol breath test at admission, or inability to abstain from alcohol during the study.

  5.Excessive consumption of tea, coffee, or other caffeinated beverages (average >8 cups/day, 1 cup = 250 mL) within 3 months prior to screening.

  6.Inability to refrain from caffeine-containing foods or beverages (e.g., coffee, strong tea, cola, chocolate) within 72 hours prior to admission or during the study, or consumption of other foods affecting drug absorption, distribution, metabolism, or excretion (e.g., dragon fruit, mango, grapefruit, pomelo, orange, starfruit, guava).

  7.Participation in another clinical trial involving drugs or devices within 3 months prior to screening, or use of investigational products prior to first admission.

  8.Vaccination (including but not limited to COVID-19, tetanus, rabies, HPV) within 2 months prior to screening.

  9.Blood donation or significant blood loss (≥400 mL) within 3 months prior to screening, transfusion or use of blood products within 3 months prior, blood loss ≥200 mL within 30 days, or plasma/aphresis donation within 7 days prior.

  10.Use of prescription drugs, over-the-counter drugs, herbal medicines, or dietary supplements within 14 days prior to screening or between screening and first admission.

  11.History of syncope related to needles or blood, difficulty with blood collection, or orthostatic hypotension.

  12.Special dietary requirements preventing adherence to a standardized diet.

  13.History of substance abuse or drug addiction, or positive test for addictive substances (methamphetamine, MDMA, THC, morphine, ketamine) on the day of admission.

  14.Pregnant or breastfeeding women, or women of childbearing potential with a positive pregnancy test.

  15.Abnormal vital signs, physical examination, laboratory tests, ECG, CT, or ultrasound deemed clinically significant by the investigator.

  16.Women using oral contraceptives within 30 days prior to screening or during the study, or long-acting estrogen/progestin injections or implants within 6 months prior to screening or during the study.

  17.Positive test for hepatitis B surface antigen, hepatitis C antibody, HIV antibody, or syphilis (Treponema pallidum) antibody.

  18.Any other condition or factor deemed by the investigator to make the participant unsuitable for the study.

  *Chronic pain is defined as persistent or recurrent pain lasting more than 3 months. Acute pain is defined as pain lasting less than 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  Cmax after single-dose administration and Cmax after the first dose in the multiple-dose group
Tmax | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  Tmax after single-dose administration and Tmax after the first dose in the multiple-dose group
AUC0-t | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  AUC0-t after single-dose administration and AUC0-t after the first dose in the multiple-dose group
AUC0-∞ | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  AUC0-∞ after single-dose administration and AUC0-∞ after the first dose in the multiple-dose group

SECONDARY OUTCOMES:
t1/2 | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  t1/2 after single-dose administration and t1/2 after the first dose in the multiple-dose group
λz | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  λz after single-dose administration and λz after the first dose in the multiple-dose group
AUC_%Extrap | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  AUC_%Extrap after single-dose administration and AUC_%Extrap after the first dose in the multiple-dose group
Css_min | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  Trough concentration at steady state (Css_min) in the multiple-dose group
Css_max | Within 60 minutes prior to dosing, and at 5, 15, 30, and 45 minutes, and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, and 12 hours post-dose.
  Peak concentration at steady state (Css_max) in the multiple-dose group
TNF-α | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Tumor Necrosis Factor-α
IFN-γ | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Interferon-γ
IL-6 | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Interleukin-6
IL-10 | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Interleukin-10
IL-17A | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Interleukin-17A
CD3+ T cell | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  CD3+ T cell subsets
CD4+ T cell | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  CD4+ T cell subsets
CD8+ T cell | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  CD8+ T cell subsets
ANA | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Antinuclear Antibody
ESR | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Erythrocyte Sedimentation Rate
CRP | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  C-Reactive Protein
Ig E | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Immunoglobulin E
Ig G | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Immunoglobulin G
Ig M | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Immunoglobulin M
Ig A | single-dose group: baseline and at Day 8 and Day 15 post-dose; multiple-dose group: baseline and at Day 35 and Day 49 post-dose.
  Immunoglobulin A

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China